CLINICAL TRIAL: NCT03889522
Title: The Influence of Non-Caloric Artificial Sweeteners on the Metabolome, Body Composition, and Glycemic Control in Youth With Type 1 Diabetes
Brief Title: The Influence of Non-Caloric Artificial Sweeteners on Youth With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Susanne Cabrera, Associate Professor, Medical College of Wisconsin
Other Study IDs: 1351723
Record Dates: First submitted 2019-02-20; First posted 2019-03-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood plasma will be used for metabolomic analyses. Samples will be stored and used until none is left.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Bioelectrical Impedance Analysis — BIA is a radiation-free and clinically accessible measure of body composition [47, 49]. An electrode is placed on the youth's extremities and they are asked to sit for 10 minutes. The youth's height and weight is manually inputted and the measure is obtained (approx. 90 seconds to complete). BIA sends a low level of electrical current through the body and measures the impedance to the current based on fat, muscle, bones providing a measure of body composition.
  Other Names: BIA
Diagnostic Test: Total Body Dual-energy X-ray Absorptiometry — The DXA total body scan provides measurements of percent body fat, lean and fat free mass throughout the body. Youth lay on a table while the machine moves around them. The process takes about 3 minutes and 20 seconds.
  Other Names: DXA
Diagnostic Test: Blood draw — Blood will be drawn to assess the following labs: HbA1c, leptin, lipid panel and comprehensive metabolic panel.

SUMMARY:
The investigators aim to further the understanding of environmental factors that may underlie variations in body composition seen in youth with Type 1 diabetes (T1D). Non-caloric artificial sweeteners, broadly consumed in many individuals with T1D, are a modifiable dietary factor that may be associated with negative health outcomes, particularly those relevant to the future risk of diabetes-related complications.

Investigators will measure body composition (the amount of fat and muscle in the body and where the fat is stored) using a bioelectrical impedance analysis machine and DEXA scanner. Blood will be drawn for the following labs: HbA1c, lipid panel, comprehensive metabolic panel and leptin. Participants will also answer questions about their diets and consumption of artificial sweeteners.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 5-17 years with a clinical diagnosis of T1D of ≥ 6 months in duration
2. BMI between the 5th and 95th percentile

Exclusion Criteria:

1. Presence of severe, active disease that requires the use of chronic medication, with the exception of well-controlled autoimmune thyroiditis/hypothyroidism or celiac disease that is well-controlled on a gluten free diet.
2. Diabetes other than T1D
3. Chronic illness known to affect glucose metabolism
4. Psychiatric impairment, with the exception of well-controlled depression or anxiety, that will affect the ability to participate in the study
5. Female participants of child-bearing age with reproductive potential must not be knowingly pregnant
6. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Youth receiving care at the Children's Hospital of Wisconsin Diabetes Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Quantify artificial sweetener consumption in youth with type 1 diabetes | Study Duration (1 year)
  To quantify artificial sweetener consumption patterns in a cohort of youth with T1D through novel food frequency questionnaires (Non-caloric artificial sweetener Food Frequency Questionnaire for Food and the Non-caloric artificial sweetener Food Frequency Questionnaire for Beverages) and bioassay
Examine the relationship between artificial sweeteners and body composition | Study Duration (1 year)
  To characterize the relationship between artificial sweetener consumption and measures of body composition, as measured by bioelectrical impedance analysis and DXA scanning, which provide information on the amount and distribution of fat and muscle in the body.
Examine the relationship between artificial sweeteners and kidney function | Study Duration (1 year)
  To determine if the level of artificial sweeteners is associated with the serum creatinine level.
Examine the relationship between artificial sweeteners and liver function | Study Duration (1 year)
  To determine if the level of artificial sweeteners is associated with serum AST and ALT levels
Examine the relationship between artificial sweeteners and lipid levels. | Study Duration (1 year)
  To characterize the relationship between artificial sweetener consumption and metabolism and the levels of fasting lipids (triglyceride level, HDL, LDL, and total cholesterol).
Examine the relationship between artificial sweeteners and metabolism. | Study Duration (1 year)
  To characterize the relationship between artificial sweetener consumption and metabolism, as measured by a leptin level.
Examine the relationship between artificial sweeteners and glycemic control | Study Duration (1 year)
  To characterize the relationship between artificial sweetener consumption and measures of glycemic control, as determined by the presence or absence of microalbuminuria.
Examine the relationship between artificial sweeteners and glycemic control | Study Duration (1 year)
  To characterize the relationship between artificial sweetener consumption and measures of glycemic control, as measured by total daily insulin dose.
Examine the relationship between artificial sweeteners and glycemic control | Study Duration (1 year)
  To characterize the relationship between artificial sweetener consumption and measures of glycemic control, as measured by the percentage of time participants are within ideal range for blood glucose levels (as measured by glucose monitors.)
Examine the relationship between artificial sweeteners and hemoglobin A1c | Study Duration (1 year)
  To characterize the relationship between artificial sweetener consumption and measures of glycemic control, as measured by serum HbA1c.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No